CLINICAL TRIAL: NCT02070315
Title: Quantitative Evaluation of Liver Disease With Liver and Kidney Elastography Using the Supersonic Imagine Aixplorer ShearWaveTM Elastography Ultrasound Machine
Brief Title: Quantitative Evaluation of the Progression of Liver Disease, Using ShearWaveTM
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 012-011
Record Dates: First submitted 2013-01-08; First posted 2014-02-25 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2022-08

CONDITIONS: Liver Disease; Heart Failure
Keywords: heart failure; liver failure; post liver transplant
MeSH Terms: conditions — Liver Diseases; Heart Failure; Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Liver biopsy for the assessment of fibrosis has multiple limitations. Liver ShearWaveTM Elastography may provide a non-invasive, fast, and reproducible alternative for the quantitative assessment of liver fibrosis.

DETAILED DESCRIPTION:
To obtain a quantitative evaluation of the progression of liver disease, using ShearWaveTM Elastography measurements obtained with the Supersonic Imagine Aixplorer ultrasound machine.

To compare the glomerular filtration rate and the quantitative evaluation of the progression of renal disease, using ShearWaveTM Elastography measurements obtained with the Supersonic Imagine Aixplorer ultrasound machine in post-liver transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females over the age of 18
* Patients of Liver Consultant's of Texas Dallas office, with chronic liver disease or liver transplant patient seen in Liver Transplant Clinic
* Patients diagnosed with heart failure

Exclusion Criteria:

- Any person unable to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants will be from Liver Consultants of Texas patient population
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2012-02; Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Shearwave Elastography Ultrasound | 1 day
  Patients will have a scan performed at their regularly scheduled clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: James Trotter, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided